CLINICAL TRIAL: NCT03625674
Title: Impact of Stigma on Compliance to Medication in Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, professor, chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJYYXHNK-003
Record Dates: First submitted 2018-07-24; First posted 2018-08-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-08

CONDITIONS: Functional Gastrointestinal Disorders; Adherence, Patient
MeSH Terms: conditions — Gastrointestinal Diseases; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- psychological and GI mechanisms (Other): The patients in Group 1 were told that: GI symptoms in FD are attributable to both psychological and GI mechanisms. Psychoactive medicine relieves FD symptoms through both psychological and GI mechanisms.
  Interventions: Behavioral: explanation when prescribing psychoactive medicine
- psychological mechanism (Other): The patients in Group 2 were told that: GI symptoms in FD are attributable to psychological mechanisms. Psychoactive medicine relieves FD symptoms through psychological mechanisms.
  Interventions: Behavioral: explanation when prescribing psychoactive medicine
- GI mechanism (Other): The patients in Group 3 were told that: GI symptoms in FD are attributable to GI mechanisms. Psychoactive medicine relieves FD symptoms through GI mechanisms.
  Interventions: Behavioral: explanation when prescribing psychoactive medicine
- no explanation (Other): The patients in Group 4 were not explained with the detailed mechanism of FD and psychoactive medicine
  Interventions: Behavioral: explanation when prescribing psychoactive medicine

INTERVENTIONS:
Behavioral: explanation when prescribing psychoactive medicine — explanation of the pathogenesis of FD and the mechanism of psychoactive medicine

SUMMARY:
To date, no study exists that evaluates whether functional dyspepsia patients experience stigma and how stigma may influence adherence. Thus, the investigators aim to evaluate the relationship between functional dyspepsia and stigma, and explore possible ways to improve treatment adherence.

DETAILED DESCRIPTION:
Due to the functional but refractory nature of functional gastrointestinal diseases (FGIDs), large number of patients who suffer from FGIDs may not be able to fully understand their diagnosis, especially when they were told that they had no organic disease and their symptoms had a psychosomatic origin rather than a gastrointestinal one. Moreover, subjects with FGIDs have concerns and negative perceptions about medications, particularly in the presence of psychiatric comorbidity. Fearing of being labeled as insane or incapability, many patients with psychosomatic symptoms choose to conceal their illness to family, colleagues and doctors. These factors may affect willingness to initiate neuromodulator regimens and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old;
* met the ROME IV criteria for FD;
* absence of abnormalities in physical examination, laboratory tests (including a routine blood test, blood glucose, and liver function examination), abdominal ultrasonography and upper GI endoscopy within 6 months;
* absence of H. pylori infection;
* Generalized Anxiety Disorder Scale (GAD-7) ≥ 1 or Patient Health Questionnaire Depression Scale (PHQ-9) ≥ 5

Exclusion Criteria:

* any evidence of organic digestive diseases;
* other FGIDs such as IBS;
* severe psychological symptoms with GAD-7 ≥ 11 or PHQ-9 ≥15;
* pregnancy or breastfeeding; recent myocardial infarction or cardiac arrhythmias;
* previous gastric surgery;
* use of PPIs, psychoactive drugs or other drugs that might affect gastric function within 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
compliance of psychoactive medicine | week8
  Compliance is assessed by the medication possession ratio(MPR). The MPR is often defined as the sum of the days' supply of medication divided by the number of days between the first fill and the last refill plus the days' supply of the last refill. This calculation usually results in a ratio less than 1.0 if there are lapses in prescription refilling.

SECONDARY OUTCOMES:
stigma scale | week 0
  Stigma is assessed by internalized stigma of mental illness (ISMI) scale and perceived stigma (PSS) scale adapted for FD. The ISMI is a 29-item self-report questionnaire with items ranked on a 4-point Likert Scale (strongly disagree = 1 to strongly agree = 4 points). An optional fifth subscale for stigma resistance was not used in this study. Higher scores indicate greater internalized stigma: scores ≤ 2 would be labeled as 'minimal stigma', scores 2 - 2.5 were labeled as 'mild stigma', scores 2.5 - 3 were labeled as 'moderate stigma' , scores > 3 were labeled as 'severe stigma'. The PSS is a 10-item questionnaire with items ranked on a 5-point Likert Scale (seldom = 1 to always = 5 points). Higher scores indicate greater levels of perceived stigma.
dyspepsia symptom score | week 2, week 4, week 6, week8
  Participates' dyspeptic symptoms is assessed using the Leeds dyspepsia scale( LDQ), which is a reliable, valid and responsive outcome measure for quantifying the frequency and severity of dyspepsia symptoms. The LDQ contains eight items about epigastric pain, retro-sternal pain, regurgitation, nausea, vomiting, belching, early satiety and dysphagia with six grades for each item. LDQ scores of 0 - 4 were classified as very mild dyspepsia, 4 - 8 as mild dyspepsia, 9 -15 as moderate dyspepsia, and > 15 as severe or very severe dyspepsia.
anxiety symptom scores | week 2, week 4, week 6, week8
  The anxiety condition is evaluated with the Generalized Anxiety Disorder Scale (GAD-7). The GAD-7 has good performance characteristics in screening generalized anxiety disorder and are feasible for use. The GAD-7 consists of 7 items on a four-point (0 - 3) scale. Scores of 0 to 4 can be regarded as absent of generalized anxiety disorder, , scores of 5 to 9 are suggestive of mild, scores of 10 to 14 indicate moderate, and scores of 15 or higher indicate severe generalized anxiety disorder.
depression symptom scores | week 2, week 4, week 6, week8
  The depression condition is evaluated with the Patient Health Questionnaire Depression Scale (PHQ-9). The PHQ-9 is a 10-item questionnaire and has been proven to be a valid and efficient tool for screening depression. Scores of 0 to 4 can be regarded as none or minimal depression, scores of 5-9 as mild, scores of 10 to 14 are suggestive of moderate, scores of 15-19 as moderately severe, and scores of 20 or higher indicate severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- RenJiH, Shanghai, China

REFERENCES:
- [Derived] Yan XJ, Luo QQ, Qiu HY, Ji CF, Chen SL. The impact of stigma on medication adherence in patients with functional dyspepsia. Neurogastroenterol Motil. 2021 Feb;33(2):e13956. doi: 10.1111/nmo.13956. Epub 2020 Jul 27. PMID 33184967